CLINICAL TRIAL: NCT04829162
Title: Weight Stigma by Association Among Parents of Children With Obesity
Brief Title: Weight Stigma by Association in Parent-Child Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, A. Janet Tomiyama, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Parent Stigma
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Childhood Obesity; Obesity
Keywords: childhood obesity; weight stigma by association; parenting
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Adiposity; Nuclear Family

STUDY DESIGN:
Intervention Model Description: We conducted a 2 (parent with versus without obesity) x 2 (child with versus without obesity) x 2 (daughter versus son) x 2 (mother versus father) between-subjects experiment. Participants were randomly assigned to one of 16 conditions. However, only five a priori hypotheses were tested.
Who Masked: Investigator
Masking Description: Investigator was blind to condition throughout data accrual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Mother with obesity, daughter with obesity (Experimental): Image of a mother with obesity and a daughter with obesity.
  Interventions: Other: Mother with obesity, daughter with obesity
- Mother with obesity, daughter without obesity (Experimental): Image of a mother with obesity and a daughter without obesity.
  Interventions: Other: Mother with obesity, daughter without obesity
- Mother without obesity, daughter with obesity (Experimental): Image of a mother without obesity and a daughter with obesity.
  Interventions: Other: Mother without obesity, daughter with obesity
- Mother without obesity, daughter without obesity (Experimental): Image of a mother without obesity and a daughter without obesity.
  Interventions: Other: Mother without obesity, daughter without obesity
- Mother with obesity, son with obesity (Experimental): Image of a mother with obesity and a son with obesity.
  Interventions: Other: Mother with obesity, son with obesity
- Mother with obesity, son without obesity (Experimental): Image of a mother with obesity and a son without obesity.
  Interventions: Other: Mother with obesity, son without obesity
- Mother without obesity, son with obesity (Experimental): Image of a mother without obesity and a son with obesity.
  Interventions: Other: Mother without obesity, son with obesity
- Mother without obesity, son without obesity (Experimental): Image of a mother without obesity and a son without obesity.
  Interventions: Other: Mother without obesity, son without obesity
- Father with obesity, daughter with obesity (Experimental): Image of a father with obesity and a daughter with obesity.
  Interventions: Other: Father with obesity, daughter with obesity
- Father with obesity, daughter without obesity (Experimental): Image of a father with obesity and a daughter without obesity.
  Interventions: Other: Father with obesity, daughter without obesity
- Father without obesity, daughter with obesity (Experimental): Image of a father without obesity and a daughter with obesity.
  Interventions: Other: Father without obesity, daughter with obesity
- Father without obesity, daughter without obesity (Experimental): Image of a father without obesity and a daughter without obesity.
  Interventions: Other: Father without obesity, daughter without obesity
- Father with obesity, son with obesity (Experimental): Image of a father with obesity and a son with obesity.
  Interventions: Other: Father with obesity, son with obesity
- Father with obesity, son without obesity (Experimental): Image of a father with obesity and a son without obesity.
  Interventions: Other: Father with obesity, son without obesity
- Father without obesity, son with obesity (Experimental): Image of a father without obesity and a son with obesity.
  Interventions: Other: Father without obesity, son with obesity
- Father without obesity, son without obesity (Experimental): Image of a father without obesity and a son without obesity.
  Interventions: Other: Father without obesity, son without obesity

INTERVENTIONS:
Other: Mother with obesity, daughter with obesity — Participants in this group were shown an image of a mother with obesity and a daughter with obesity.
  Arms: Mother with obesity, daughter with obesity
Other: Mother with obesity, daughter without obesity — Participants in this group were shown an image of a mother with obesity and a daughter without obesity.
  Arms: Mother with obesity, daughter without obesity
Other: Mother without obesity, daughter with obesity — Participants in this group were shown an image of a mother without obesity and a daughter with obesity.
  Arms: Mother without obesity, daughter with obesity
Other: Mother without obesity, daughter without obesity — Participants in this group were shown an image of a mother without obesity and a daughter without obesity.
  Arms: Mother without obesity, daughter without obesity
Other: Mother with obesity, son with obesity — Participants in this group were shown an image of a mother with obesity and a son with obesity.
  Arms: Mother with obesity, son with obesity
Other: Mother with obesity, son without obesity — Participants in this group were shown an image of a mother with obesity and a son without obesity.
  Arms: Mother with obesity, son without obesity
Other: Mother without obesity, son with obesity — Participants in this group were shown an image of a mother without obesity and a son with obesity.
  Arms: Mother without obesity, son with obesity
Other: Mother without obesity, son without obesity — Participants in this group were shown an image of a mother without obesity and a son without obesity.
  Arms: Mother without obesity, son without obesity
Other: Father with obesity, daughter with obesity — Participants in this group were shown an image of a father with obesity and a daughter with obesity.
  Arms: Father with obesity, daughter with obesity
Other: Father with obesity, daughter without obesity — Participants in this group were shown an image of a father with obesity and a daughter without obesity.
  Arms: Father with obesity, daughter without obesity
Other: Father without obesity, daughter with obesity — Participants in this group were shown an image of a father without obesity and a daughter with obesity.
  Arms: Father without obesity, daughter with obesity
Other: Father without obesity, daughter without obesity — Participants in this group were shown an image of a father without obesity and a daughter without obesity.
  Arms: Father without obesity, daughter without obesity
Other: Father with obesity, son with obesity — Participants in this group were shown an image of a father with obesity and a son with obesity.
  Arms: Father with obesity, son with obesity
Other: Father with obesity, son without obesity — Participants in this group were shown an image of a father with obesity and a son without obesity.
  Arms: Father with obesity, son without obesity
Other: Father without obesity, son with obesity — Participants in this group were shown an image of a father without obesity and a son with obesity.
  Arms: Father without obesity, son with obesity
Other: Father without obesity, son without obesity — Participants in this group were shown an image of a father without obesity and a son without obesity.
  Arms: Father without obesity, son without obesity

SUMMARY:
Parents of children with obesity report feeling blamed for their children's weight and reluctant to seek pediatric care after stigmatizing experiences. This "weight stigma by association" may have direct consequences for parents, children, and the parent-child relationship. The present study builds on qualitative evidence to experimentally test weight stigma and weight stigma by association in a parent-child relationship using a large, community-based sample. In an experiment conducted via an online survey, participants were randomly assigned to view a picture of a parent-child dyad, for which parent and child's gender (male vs. female) and weight status (with obesity vs. without obesity) were manipulated. Participants read identical general parenting descriptions that adhered to American Academy of Pediatrics parenting recommendations, then rated the parent's effectiveness, helpfulness, and caring.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age

Exclusion Criteria:

* Standard exclusion criteria were duplicate IP addresses, response times < 60s or > 3600s (the allotted time to complete the survey), or failure to complete the parenting questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1973 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Parenting evaluation | 1 day
  Participants responded to the prompt, "To what extent do you perceive the parenting approach to be effective/helpful/caring?" and rated the characteristic on a 5-point Likert scale (1 = Not at all, 5 = Very).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No